CLINICAL TRIAL: NCT05277506
Title: Smile Arc Assessment in Orthodontic Patients Following Smile Arc Protection Versus MBT Placement Guide Bonding Strategies: A Randomized Clinical Trial.
Brief Title: Smile Arc Assessment in Orthodontic Patients Following Smile Arc Protection VS MBT Placement Guide Bonding Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Hamza Hassan Saleh, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORTH 3-3-3
Record Dates: First submitted 2022-02-18; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smile arc protection bonding strategy group (Experimental): female patients with mild crowding will recieve orthodontic brackets bonding using smile arc protection bonding strategy
  Interventions: Device: 18 inch slot MBT orthodontic brackets bonded using smile arc protection bonding strategy
- MBT placement guide group (Active Comparator): female patients with mild crowding will recieve orthodontic brackets bonding using MBT placement guide
  Interventions: Device: 18 inch slot MBT orthodontic brackets boned using MBT placement guide

INTERVENTIONS:
Device: 18 inch slot MBT orthodontic brackets bonded using smile arc protection bonding strategy — female patients with mild crowding will recieve orthodontic brackets bonding using smile arc protection bonding strategy
  Arms: smile arc protection bonding strategy group
Device: 18 inch slot MBT orthodontic brackets boned using MBT placement guide — female patients with mild crowding will recieve orthodontic brackets bonding using MBT placement guide bonding strategy
  Arms: MBT placement guide group

SUMMARY:
The study will be performed on human subjects undergoing orthodontic treatment to correct mild crowding with both techniques enhancing the final smile characteristics of the patients.

DETAILED DESCRIPTION:
The study concisits of two groups, the intervention group entails performing bonding of orthodontic brackets following smile arc protection bonding strategy while the control group entails performing bonding using the MBT placement guide and comparing the final smile outcomes after reaching steel archwires for both groups using customized questionnaires for orthodontists and laypersons.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* no/mild/moderate crowding or spacing
* non-extraction treatment decision with non-extraction profile
* adults age 16-30 years
* full permanent dentition including fully erupted 7s not necessarily 8s
* good oral hygiene.

Exclusion Criteria:

* severe crowding
* cleft lip and palate/syndromic patients
* bad oral hygiene
* unerupted or partially erupted 7s
* extracted or missing teeth

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female patients 16-30 years
Enrollment: 22 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
smile arc assessment by orthodontists | 6 months follow up
  subjective assessment of the beauty of the smile using close up photographs and questionnaires filled by orthodontists and graded scale from 0-10

SECONDARY OUTCOMES:
smile arc analysis using frontal extraoral photographs of the posed smile | 6 months follow up
  analysis in millimeters for anthropometric measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Faculty of Dentistry., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No